CLINICAL TRIAL: NCT05780320
Title: A Pharmaco-surgical Approach to Reduce Postoperative Atrial Fibrillation After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Asishana A Osho, Assistant Professor of Surgery, Massachusetts General Hospital
Other Study IDs: 2004P001528
Record Dates: First submitted 2023-02-28; First posted 2023-03-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Postoperative atrial fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pharmaco-Surgical Arm
  Interventions: Other: Prophylactic amiodarone and posterior pericardiotomy
- Standard of Care Arm

INTERVENTIONS:
Other: Prophylactic amiodarone and posterior pericardiotomy — Patients after the implementation of the protocol receive postoperative prophylactic amiodarone and a posterior pericardiotomy.
  The amiodarone regimen consists of amiodarone 1mg/min x 10 hours (600 mg total) via central line upon arrival to the intensive care unit followed by 400 mg PO BID on postoperative days 1 and 2 followed by 200 mg PO BID on postoperative days 3 and 4 or until discharge, whichever occurs first.
  The posterior pericardiotomy occurs during the cardiac procedure.
  Groups: Pharmaco-Surgical Arm

SUMMARY:
Postoperative atrial fibrillation (POAF) is a common complication following cardiac surgery with an estimated incidence around 35%. It has been found to be an independent predictor of 30-day and 6-month mortality, stroke, renal failure, respiratory failure, and need for permanent pacemaker among others. Previous studies including meta-analyses demonstrate a protective benefit of prophylactic amiodarone to decrease the risk of POAF. However, this has not been widely adopted, and recent society guidelines only give prophylactic amiodarone a Class IIA recommendation, citing risk of amiodarone-related toxicity and hypotension as reasons for the Class IIA recommendation. A meta-analysis comparing cumulative doses of amiodarone found that moderate to higher doses of amiodarone have a marginally increased benefit in reducing the incidence of postoperative atrial fibrillation over lower doses; however, the study did not assess risk of complications stratified by cumulative doses, which has been previously described. Finally, a recent meta-analysis showed that a posterior pericardiotomy was highly effective at reducing postoperative atrial fibrillation. Consequently, the investigators' institution has adopted a pharmaco-surgical approach (prophylactic amiodarone and posterior pericardiotomy) in an effort to reduce postoperative atrial fibrillation after coronary artery bypass cardiac surgery for all patients who meet inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative normal sinus rhythm
* Procedures:
* CABG
* CABG + concomitant valve or aortic replacement/repair

Exclusion Criteria:

* Emergent operation

Procedures:

* MAZE or PVI performed
* Isolated valve replacement or repair
* Isolated aortic procedures
* Heart transplant
* Lung transplant Pre-existing atrial arrhythmias Pre-operative amiodarone use Contraindications to amiodarone use
* PR interval > 240 ms
* 2nd or 3rd degree heart block
* QTc > 550ms
* 2nd or 3rd degree heart block
* Liver impairment (INR > 1.7, AST/ALT > 2x normal)
* Uncontrolled hypothyroidism/hyperthyroidism
* Interstitial lung disease
* Allergy to amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all patients undergoing coronary artery bypass cardiac surgery at the Massachusetts General Hospital who meets the above criteria.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | Prior to patient discharge or within 30 days after surgery.
  At least 1 minute duration detected by continuous telemetry or 12-lead electrocardiogram.

SECONDARY OUTCOMES:
Operative mortality | Either in-hospital death or death within 30 days of discharge
  Operative mortality as defined by either in-hospital death or death within 30 days of discharge.
Stroke | Either in-hospital or within 30 days of procedure
  Characterized by deficits lasting > 24 hours and/or imaging findings of infarction
Transient ischemic attack | Either in-hospital or within 30 days of procedure
  Characterized by examination findings lasting < 24 hours without associated imaging findings
Initiation of systemic anticoagulation | Either in-hospital or within 30 days of procedure
  New indication of systemic anticoagulation for stroke prophylaxis due to atrial fibrillation
Persistence of atrial fibrillation at discharge | At postoperative surgical visit (around 4-6 weeks)
  Atrial fibrillation as diagnosed by final ECG
Postoperative hospital length of stay | Up to 90 days
  The postoperative length of stay will be calculated starting from the end of the procedure to time of discharge
Readmission | Within 30 days of procedure
  Rates of hospital readmission will be estimated for patients in each of the study intervention groups. Readmissions will be counted in this calculation if patients are admitted to the hospital. Emergency room visits without admission and outpatient visits will not count toward this calculation of readmission rates.
Symptomatic bradycardia | Either in-hospital or within 30 days of procedure
  Symptomatic bradycardia (HR < 55 bpm) requiring intervention
Number of patients with Amiodarone-related pulmonary toxicity | Either in-hospital or within 30 days of procedure
  Clinical diagnosis of amiodarone-related pulmonary toxicity that uses a combination of x-ray findings consistent with known amiodarone-related pulmonary toxicity and clinical findings including shortness of breath, non-productive cough, and other diagnoses have been excluded.
Postoperative pleural effusions requiring intervention | Either in-hospital or within 30 days of procedure
  Postoperative pleural effusions requiring interventions including thoracostomy drainage or surgical drainage

CONTACTS AND LOCATIONS:
Overall Officials: Asishana A Osho, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenberg JW, Lancaster TS, Schuessler RB, Melby SJ. Postoperative atrial fibrillation following cardiac surgery: a persistent complication. Eur J Cardiothorac Surg. 2017 Oct 1;52(4):665-672. doi: 10.1093/ejcts/ezx039. PMID 28369234
- [Background] Arsenault KA, Yusuf AM, Crystal E, Healey JS, Morillo CA, Nair GM, Whitlock RP. Interventions for preventing post-operative atrial fibrillation in patients undergoing heart surgery. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003611. doi: 10.1002/14651858.CD003611.pub3. PMID 23440790
- [Background] Chatterjee S, Sardar P, Mukherjee D, Lichstein E, Aikat S. Timing and route of amiodarone for prevention of postoperative atrial fibrillation after cardiac surgery: a network regression meta-analysis. Pacing Clin Electrophysiol. 2013 Aug;36(8):1017-23. doi: 10.1111/pace.12140. Epub 2013 Apr 29. PMID 23627761
- [Background] Buckley MS, Nolan PE Jr, Slack MK, Tisdale JE, Hilleman DE, Copeland JG. Amiodarone prophylaxis for atrial fibrillation after cardiac surgery: meta-analysis of dose response and timing of initiation. Pharmacotherapy. 2007 Mar;27(3):360-8. doi: 10.1592/phco.27.3.360. PMID 17316148
- [Background] Colunga Biancatelli RM, Congedo V, Calvosa L, Ciacciarelli M, Polidoro A, Iuliano L. Adverse reactions of Amiodarone. J Geriatr Cardiol. 2019 Jul;16(7):552-566. doi: 10.11909/j.issn.1671-5411.2019.07.004. PMID 31447894
- [Background] Orr CF, Ahlskog JE. Frequency, characteristics, and risk factors for amiodarone neurotoxicity. Arch Neurol. 2009 Jul;66(7):865-9. doi: 10.1001/archneurol.2009.96. PMID 19597088
- [Background] Wolkove N, Baltzan M. Amiodarone pulmonary toxicity. Can Respir J. 2009 Mar-Apr;16(2):43-8. doi: 10.1155/2009/282540. PMID 19399307
- [Background] Gaudino M, Sanna T, Ballman KV, Robinson NB, Hameed I, Audisio K, Rahouma M, Di Franco A, Soletti GJ, Lau C, Rong LQ, Massetti M, Gillinov M, Ad N, Voisine P, DiMaio JM, Chikwe J, Fremes SE, Crea F, Puskas JD, Girardi L; PALACS Investigators. Posterior left pericardiotomy for the prevention of atrial fibrillation after cardiac surgery: an adaptive, single-centre, single-blind, randomised, controlled trial. Lancet. 2021 Dec 4;398(10316):2075-2083. doi: 10.1016/S0140-6736(21)02490-9. Epub 2021 Nov 14. PMID 34788640